CLINICAL TRIAL: NCT06176313
Title: Investigation of the Effects of Training Given to Cope With Premenstrual Syndrome and Mandala Activity on Premenstrual Symptoms
Brief Title: Effects of Training Given to Cope With Premenstrual Syndrome and Mandala Activity on Premenstrual Symptoms
Acronym: MANDALA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Merve SEZER YILDIZ, Phd.Student and Research Assistant, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: merve-sezer-yildiz-001
Record Dates: First submitted 2023-12-01; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Premenstrual Syndrome
Keywords: premenstrual syndrome; mandala; education; premenstrual symptoms
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Coping Skills; Control Groups

STUDY DESIGN:
Intervention Model Description: The research employs a pre-test post-test control group design with a randomized controlled semi-experimental approach to determine the impact of education provided for coping with premenstrual syndrome and Mandala activity on premenstrual symptoms.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be performed by an investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mandala (Experimental)
  Interventions: Other: Mandala Group
- Coping with Premenstrual Symptoms Education Group (Experimental)
  Interventions: Other: Coping with Premenstrual Symptoms Education Group
- Control Group (Experimental)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Mandala Group — The Mandala activity lasts approximately 60 minutes.
  • A calm environment is provided during the Mandala activity, and participants are ensured not to be disturbed by external stimuli or individuals unless they request assistance.
  Each student's last menstrual date is recorded in an Excel table.
  * Two days before the intervention day, students will be contacted and invited to participate in the study.
  * Monitoring each student's menstrual cycle, the Mandala activity intervention is scheduled during the late luteal phase of each student's menstrual cycle. The intervention is planned within the 5 days before the expected start of menstrual bleeding on days and hours convenient for the student's class schedule.
  * After each session, on the 4th day of the expected menstrual bleeding, students are subjected to PMSÖ.
  * On the 4th day of the 4th menstrual period bleeding, the research will be concluded by applying the post-test with PMSÖ to the students."
  Arms: mandala
Other: Coping with Premenstrual Symptoms Education Group — The education will be conducted through face-to-face interviews in the master's course classroom at the Faculty of Health Sciences at Bilecik Şeyh Edebali University. The education was conducted using PowerPoint presentations projected onto a white smartboard.
  * One month after the completion of the education, a 1st Reminder training will be provided in the master's course classroom within the Faculty of Health Sciences at Bilecik Şeyh Edebali University, using the face-to-face interview method.
  * One month after the 1st Reminder training, a 2nd Reminder training will be provided in the master's course classroom within the Faculty of Health Sciences at Bilecik Şeyh Edebali University, using the face-to-face interview method.
  * On the 4th day of the 4th menstrual period bleeding, the research will be concluded by applying the post-test with PMSÖ to the students.
  Arms: Coping with Premenstrual Symptoms Education Group
Other: Control Group — No intervention will be applied to the control group throughout the research. However, students in this group who cope with premenstrual syndrome using medication or non-medication methods will be monitored during the three-month menstrual cycle.
  Each student's menstrual cycle in the control group has been recorded in the Excel table. The estimated end of menstruation for each student has been noted.
  * At the estimated end of menstruation, the researcher contacts the students in the control group to inquire whether they have used any medication or non-medication methods to cope with premenstrual syndrome.
  * Those who use medication or non-medication methods to reduce premenstrual symptoms are excluded from the study.
  * On the 4th day of the 4th menstrual period bleeding, the post-test with PMSÖ will be applied to the students."
  Arms: Control Group

SUMMARY:
The research employs a pre-test post-test control group design with a randomized controlled semi-experimental approach to determine the impact of education provided for coping with premenstrual syndrome and Mandala activity on premenstrual symptoms.

Research Hypotheses:

H01: Mandala activity is not effective in reducing premenstrual symptoms.

H02: Education provided for coping with premenstrual syndrome is not effective in reducing premenstrual symptoms.

H13: Mandala activity is effective in reducing premenstrual symptoms.

H14: Education provided for coping with premenstrual syndrome is effective in reducing premenstrual symptoms.

H15: Mandala activity is more effective than education provided for coping with premenstrual syndrome in reducing premenstrual symptoms among students with PMS.

Research Groups: Mandala Group, Coping with Premenstrual Symptoms Education Group, and Control Group.

DETAILED DESCRIPTION:
In the conducted international and national literature review, it was observed that various methods are utilized in the management of PMS. Still, no study directly examining the effectiveness of Mandala activity on PMS was found. The literature results provided under the title of Mandala indicate that the activities are predominantly focused on behavioral and psychological conditions. Considering the symptoms of PMS, it is assumed that Mandala activity may have an impact on the behavioral and psychological symptoms of PMS. The assumption of how it might affect the physical symptoms of PMS is also supported by studies indicating that art itself has a therapeutic quality and that the creative process helps individuals develop positive coping methods for the physical discomfort they experience.

The research is planned as a pre-test post-test control group design with a randomized controlled semi-experimental approach, aiming to determine the impact of education on coping with premenstrual syndrome and Mandala activity on premenstrual symptoms

Research Hypotheses:

H01: Mandala activity is not effective in reducing premenstrual symptoms.

H02: Education provided for coping with premenstrual syndrome is not effective in reducing premenstrual symptoms.

H13: Mandala activity is effective in reducing premenstrual symptoms.

H14: Education provided for coping with premenstrual syndrome is effective in reducing premenstrual symptoms.

H15: Mandala activity is more effective than education provided for coping with premenstrual syndrome in reducing premenstrual symptoms among students with PMS.

Research Groups: Mandala Group, Coping with Premenstrual Symptoms Education Group, and Control Group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25 years
* Female students enrolled in the 1st and 2nd years of the Faculty of Health Sciences PMSÖ score of 110 and above
* Regular menstruation in the last six months (between 21-35 days)
* Not using any medication or non-medication methods to cope with PMS symptoms
* Not using contraceptive pills
* Absence of any gynecological diseases (abnormal uterine bleeding, fibroids, ovarian cysts, etc.)
* No diagnosis of psychiatric illness
* Not using any psychiatric medication such as antidepressants
* Absence of any condition that may hinder Mandala drawing
* No previous experience with Mandala education
* Willingness to participate in the study
* Proficiency in speaking and understanding Turkish

Exclusion Criteria: Students who do not meet the criteria mentioned above and are not willing to participate in the study will be excluded.

-

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 90 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
the Premenstrual Syndrome Scale (PSS) for mandala pre-test | pre-test
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.
the Premenstrual Syndrome Scale (PSS) for education pre-test | pre-test
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.
the Premenstrual Syndrome Scale (PSS) for control | pre-test
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.

SECONDARY OUTCOMES:
the Premenstrual Syndrome Scale (PSS) after mandala-1 session | Four days after the first menstrual bleeding.
  Mandala sessions are conducted with students approximately 7 days before each monthly menstrual bleeding. The sessions are planned in a total of 3 sessions. Four days after each mandala session, students fill out the Premenstrual Syndrome Scale (PSS) form. The result obtained at this time represents the PSS outcome after the 1st Mandala session.
  Students who scored 110 or above on the Premenstrual Syndrome Scale (PSS) and met the inclusion criteria of the study were randomly assigned to study groups. The scores obtained by the included students on the PSS were considered as the pre-test for the study.
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.
the Premenstrual Syndrome Scale (PSS) after mandala-2 session | Four days after the second menstrual bleeding."
  Mandala sessions are conducted with students approximately 7 days before each monthly menstrual bleeding. The sessions are planned in a total of 3 sessions. Four days after each mandala session, students fill out the Premenstrual Syndrome Scale (PSS) form. The result obtained at this time represents the PSS outcome after the 2st Mandala session.
  Students who scored 110 or above on the Premenstrual Syndrome Scale (PSS) and met the inclusion criteria of the study were randomly assigned to study groups. The scores obtained by the included students on the PSS were considered as the pre-test for the study.
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.
the Premenstrual Syndrome Scale (PSS) after mandala-3 session | Four days after the third menstrual bleeding.
  Mandala sessions are conducted with students approximately 7 days before each monthly menstrual bleeding. The sessions are planned in a total of 3 sessions. Four days after each mandala session, students fill out the Premenstrual Syndrome Scale (PSS) form. The result obtained at this time represents the PSS outcome after the 3st Mandala session.
  Students who scored 110 or above on the Premenstrual Syndrome Scale (PSS) and met the inclusion criteria of the study were randomly assigned to study groups. The scores obtained by the included students on the PSS were considered as the pre-test for the study.
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.
Premenstrual Syndrome Scale (PMSS) education final test | After the third menstrual bleeding, four days later.
  Premenstrual Syndrome Scale (PMSS): PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.
Premenstrual Syndrome Scale (PMSS) control final test | After the third menstrual bleeding, four days later.
  The Premenstrual Syndrome Scale (PMSS): The PMSS consists of 44 items. The total PMSS score is obtained by summing the scores of subscales. The lowest score that can be obtained on the scale is 44, and the highest score is 220. Higher scores indicate increased severity of PMS symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Merve SEZER YILDIZ, Ph.D. Student, Principal Investigator — BİLECİK ŞEYH EDEBALİ UNİVERSITY; Özlem ÇAĞAN, Assist. Professor, Study Director — ESKİŞEHİR OSMANGAZİ UNİVERSITY
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No